CLINICAL TRIAL: NCT02421731
Title: Effectiveness of Robot-assisted Gait Training Versus Conventional Therapy on Mobility in Severely Disabled Multiple Sclerosis Patients
Brief Title: Robot-assisted Gait Training on Mobility in Severely Disabled Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Regione Emilia-Romagna (Other); Università degli Studi di Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Regionale WP3
Record Dates: First submitted 2015-01-19; First posted 2015-04-21 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Gait
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot-assisted gait training (Experimental): This group will receive rehabilitation treatment based on robot-assisted gait training.
  Interventions: Device: Robot-assisted gait training
- Conventional therapy (Active Comparator): This group will receive conventional rehabilitation therapy.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: Robot-assisted gait training — Patients will receive 12 training sessions, lasting for an hour with 30 minutes of real walking time, over 4 weeks (3 sessions/week) of RAGT. Subjects will wear a harness attached to a system to provide body weight support and they will walk on a treadmill with the help of a robotic-driven gait orthosis. The legs are guided according to a physiological gait pattern. The torque of the knee and hip drives can be adjusted from 100% to 0% for one or both legs. The speed of the treadmill can be adjusted from 0 km/h to approximately 3 km/h and body weight support from 0% to 100%. During the first session we will set these parameters according to subject characteristics and demand level. As training will progress, adjustments in the three parameters previously described will be performed.
  Arms: Robot-assisted gait training
Other: Conventional therapy — The control group will receive 12 conventional therapy sessions over 4 weeks (3 sessions/week), that will focus on gait training. Subjects will receive 1 hour of individual conventional physiotherapy for session. During the first 5-10 minutes the subjects will perform lower-limb and core stretching exercises to increase muscles flexibility; then they'll deal with lower-limb muscles strengthening exercises tailored on their baseline characteristics (10 minutes). After that, assisted over-ground walking training will be performed.
  Arms: Conventional therapy

SUMMARY:
Gait disabilities affect personal activities and quality of life of progressive multiple sclerosis (MS) patients. A robot-driven gait orthosis allowing a more effective support of walking movements and imitation of a nearly normal gait pattern during treadmill training at a higher speed has been developed and recently introduced in clinical settings. However, until now few studies evaluated the effects of Robot-Assisted Gait Training (RAGT) in a group of stroke, spinal cord injury and MS subjects.

In addition, the training-induced neural and biological changes potentially related to the mechanisms of recovery remain undefined.

The primary aims of this study are:

to test the feasibility of RAGT in a group of progressive severely disabled MS patients and to test the hypothesis that this intensive intervention could have higher benefit, compared with conventional therapy alone, in mobility improvement as assessed by the Timed 25 Foot Walk (T25FW)

The secondary aims of this study are:

to determine whether fatigue, Quality of life, balance and locomotor function are improved by RAGT; to determine whether gait training influences markers of plasticity including clinical and circulating biomarkers to search for a possible correlation between clinical outcomes and clinical and circulating biomarkers

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blinded, controlled study. Ninety-eight MS subjects will be recruited from the identification of subjects at U.O. Rehabilitative Medicine and Rare Diseases and Neuroimmune Center, IRCCS Neurosciences "Bellaria" (BO).

After evaluation of their eligibility and when obtained the informed consent, patients will be enrolled and randomized to the two groups through a randomization stratification approach. Subjects will be grouped into strata defined by the degree of impairment (e.g. using outcomes from the Expanded Disability Status Scale or EDSS) and then randomized separately within each stratum according to a block randomization and will be assigned to one of the two treatment groups:

1. robot-assisted gait training (experimental group)
2. conventional therapy (control group)

Robot-assisted gait training:

Patients will receive 12 training sessions over 4 weeks (3 sessions/week) of RAGT. During these sessions subjects will wear a harness attached to a system to provide body weight support and they will walk on a treadmill with the help of a robotic-driven gait orthosis. The legs are guided according to a physiological gait pattern. The torque of the knee and hip drives can be adjusted from 100% to 0% for one or both legs. The speed of the treadmill can be adjusted from 0 km/h to approximately 3 km/h and body weight support from 0% to 100%. During the first session we will set these training parameters according to subject characteristics and demand level. As training will progress, adjustments in the assistance provided by the driven-gait orthosis, the amount of body weight support and treadmill speed will be performed. Training sessions will last for an hour with 30 minutes of real walking time, because subject set-up in the device take approximately 30 minutes.

Conventional therapy:

The control group will receive 12 conventional therapy sessions over 4 weeks (3 sessions/week), that will focus on gait training. Subjects will receive 1 hour of individual conventional physiotherapy for session. During the first 5-10 minutes the subjects will perform lower-limb and core stretching exercises to increase muscles flexibility; then they'll deal with lower-limb muscles strengthening exercises tailored on their baseline characteristics (10 minutes). After that, assisted over-ground walking training will be performed.

Outcome measures Outcome measures will be assessed a week before the treatment initiation (T0), after two weeks (T1), after 4 weeks (T2) and at 3 months follow-up (T3). Personnel blinded to the treatment will assess the effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* severe gait impairments defined as EDSS 6-7
* lack of EDSS worsening in the last 3 months

Exclusion Criteria:

* neurologic conditions in addition to MS that may affect motor function and other medical conditions likely to interfere with the ability to safely complete the study protocol
* impaired cognitive functioning: score less than 24 on the Mini Mental State Examination
* spasticity (Ashworth scale >3) or contractures that may limit range of motion or function
* changes in disease modifying drug therapy or in any other confounding factor during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Timed 25 Foot Walk | weeks: 0,2,4,16
  The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet (7.62m) as quickly as possible, but safely, using the prescribed assistive devices.

SECONDARY OUTCOMES:
Six-Minute Walking Test | weeks: 0,2,4,16
  The walking endurance is measured with the Six-Minute Walking Test. This test, first validated in subjects with cardio-pulmonary problems, is considered a feasible, reproducible and reliable measure also in MS. Subjects are instructed to walk up and down as far as possible a 22m walkway in six minutes without encouragement, with the possibility to slow down and rest if necessary.
Berg Balance Scale | weeks: 0,2,4,16
  This is an assessment scale of ability to maintain balance, or statically or while performing functional movement, including 14 observable tasks common to everyday life measured on a 5 point ordinal scale.
Up and Go Test | weeks: 0,2,4,16
  Subjects will be given verbal instruction to stand up from a chair, walk 3 meters, cross a line marked on the floor, turn around, walk back, and sit down. A study staff member will guard the subject during the test. Subjects will perform 3 trials and the time it takes to perform each trial will be recorded with a stopwatch.
Fatigue Severity Scale | weeks: 0,2,4,16
  The Fatigue Severity Scale is a method of evaluating fatigue in MS and other conditions. Essentially, the Fatigue Severity Scale consists of answering a short questionnaire that requires the subject to to read each statement and rate his or her own level of fatigue from 1 to 7, depending on how appropriate they felt the statement applied to them over the preceding week.
Modified Ashworth Scale | weeks: 0,2,4,16
  This is a 6-point measure of spasticity. We will assess the spasticity at the hip, knee and ankle (flexors and extensors muscles).
Short-Form 36 | weeks: 0,2,4,16
  This is an assessment tool of quality of life.
Haemodynamic measurements | weeks: 0,2,4,16
  Doppler venous flow volume measurement, with evaluation of the thoracic pump; postural control of cerebral venous return assessed by plethysmography5; venous haemodynamics insufficiency severity score will be also evaluated and calculated.
Metabolic measurements by Near infrared spectroscopy | weeks: 0,2,4,16
  Near InfraRed Spectroscopy (NIRS) is a noninvasive, portable technique for ambulatory or remote monitoring of human motor-cortex oxygenation changes in response to motor tasks. Patients will walk on the treadmill at a speed of 0.2 km/h assisted by personnel and with partial body weight support, performing 4 short tasks (30 seconds of walking) alternated by rest periods (30 seconds).
Circulating biomarkers | weeks: 0,2,4,16
  blood biomarker levels modifications

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Principal Investigator — Ferrara Rehabilitation Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Italy

REFERENCES:
- [Derived] Manfredini F, Straudi S, Lamberti N, Patergnani S, Tisato V, Secchiero P, Bernardi F, Ziliotto N, Marchetti G, Basaglia N, Bonora M, Pinton P. Rehabilitation Improves Mitochondrial Energetics in Progressive Multiple Sclerosis: The Significant Role of Robot-Assisted Gait Training and of the Personalized Intensity. Diagnostics (Basel). 2020 Oct 17;10(10):834. doi: 10.3390/diagnostics10100834. PMID 33080806
- [Derived] Straudi S, Manfredini F, Lamberti N, Martinuzzi C, Maietti E, Basaglia N. Robot-assisted gait training is not superior to intensive overground walking in multiple sclerosis with severe disability (the RAGTIME study): A randomized controlled trial. Mult Scler. 2020 May;26(6):716-724. doi: 10.1177/1352458519833901. Epub 2019 Mar 4. PMID 30829117
- [Derived] Straudi S, Manfredini F, Lamberti N, Zamboni P, Bernardi F, Marchetti G, Pinton P, Bonora M, Secchiero P, Tisato V, Volpato S, Basaglia N. The effectiveness of Robot-Assisted Gait Training versus conventional therapy on mobility in severely disabled progressIve MultiplE sclerosis patients (RAGTIME): study protocol for a randomized controlled trial. Trials. 2017 Feb 27;18(1):88. doi: 10.1186/s13063-017-1838-2. PMID 28241776